CLINICAL TRIAL: NCT00578318
Title: Treatment Engagement in Psychiatric Clinical Research and Care for Depressed African American Adolescents
Brief Title: African American Knowledge Optimized for Mindfully Healthy Adolescents
Acronym: AAKOMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Alfiee Breland-Noble, Assistant Professor, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00006780 (9065); 1K01MH073814-01A1 (NIH); 5K01MH073814-02 (NIH); 5K01MH073814-03 (NIH)
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Results first posted 2013-05-17 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motivational Interviewing Active (Experimental): Patients received a stepped progression of talk based treatment utilizing Motivational Interviewing as the basis.
  Interventions: Behavioral: Motivational Interviewing Active
- Delayed Control (Active Comparator): Patients received Treatment as usual (TAU) (i.e. no specific intervention and supportive check-ins from the study staff)
  Interventions: Behavioral: Motivational Interviewing Active

INTERVENTIONS:
Behavioral: Motivational Interviewing Active — Patients received 2 sessions of an in-person talk based intervention utilizing culturally relevant Motivational Interviewing.

SUMMARY:
The purpose of this study was to better understand how African American families identify and treat emotional and behavioral concerns associated with depression in their adolescent youth. The goals of the study included (a) identifying factors associated with participation in psychiatric research and treatment and (b) developing an intervention to increase participation in psychiatric research and treatment.

DETAILED DESCRIPTION:
The aim of this study was to obtain an in-depth understanding of African Americans' perceptions of barriers to adolescent and family engagement in psychiatric treatment and research utilizing a mixed methods approach in two Phases. Phase I consisted of data collected via surveys, focus groups and individual interviews with African American adults and youth. The data generated in Phase I provided a foundation for the domains incorporated into manual development and therapist training procedures of the subsequent intervention phase of the project (Phase II).

After the research team developed the depression treatment engagement intervention, the intervention was pilot tested in a sample of depressed African American youth and families (Phase II)

ELIGIBILITY:
Inclusion Criteria:

* Persons who self-identify as Black or African American
* Adolescents aged 11 to 17 at the time of recruitment
* Adult parents
* Parent consent and adolescent assent
* Demonstrated cognitive ability to understand participation

Exclusion Criteria:

* Diminished capacity to participate

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2007-06; Primary Completion 2010-01 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfiee M Breland-Noble, Ph.D., Principal Investigator — Georgetown University
Locations (1):
- Duke Child and Family Study Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Breland-Noble AM, Bell C, Nicolas G. Family first: the development of an evidence-based family intervention for increasing participation in psychiatric clinical care and research in depressed African American adolescents. Fam Process. 2006 Jun;45(2):153-69. doi: 10.1111/j.1545-5300.2006.00088.x. PMID 16768016
- [Result] Breland-Noble AM, Bell CC, Burriss A, Poole HK; The AAKOMA Project Adult Advisory Board. The Significance of Strategic Community Engagement in Recruiting African American Youth & Families for Clinical Research. J Child Fam Stud. 2012 Apr 1;21(2):273-280. doi: 10.1007/s10826-011-9472-1. Epub 2011 Mar 4. PMID 22984337
- [Result] Breland-Noble AM; AAKOMA Project Adult Advisory Board. Community and treatment engagement for depressed African American youth: the AAKOMA FLOA pilot. J Clin Psychol Med Settings. 2012 Mar;19(1):41-8. doi: 10.1007/s10880-011-9281-0. PMID 22354616
- [Result] Breland-Noble AM, Bell CC, Burriss A; AAKOMA Project Adult Advisory Board. "Mama just won't accept this": adult perspectives on engaging depressed African American teens in clinical research and treatment. J Clin Psychol Med Settings. 2011 Sep;18(3):225-34. doi: 10.1007/s10880-011-9235-6. PMID 21512751
- [Result] Breland-Noble AM, Burriss A, Poole HK; AAKOMA PROJECT Adult Advisory Board. Engaging depressed African American adolescents in treatment: lessons from the AAKOMA PROJECT. J Clin Psychol. 2010 Aug;66(8):868-79. doi: 10.1002/jclp.20708. PMID 20564682
- See also: Study Website — http://www.aakomaproject.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study patients were recruited from the local community using tested, strategic community engagement procedures.
Groups:
- Motivational Interviewing Active: 2 sessions with parent/legal guardian and adolescent study patient of culturally relevant Motivational Interviewing intervention
- Delayed Control: At the conclusion of enrollment of all active patients, delayed control patients were offered opportunity to receive culturally relevant Motivational Interviewing intervention.
Period: Overall Study
Arm/Group | Motivational Interviewing Active | Delayed Control
Started | 8 | 8
Completed | 5 | 8
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivational Interviewing Active | Delayed Control | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 8 | 16
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Attendance at First Depression Treatment Appointment
Description: Patients were randomized to the intervention or a delayed control group. The primary outcome was bifurcated as yes or no to specify whether or not the patient attended the first available depression treatment appointment scheduled after he/she completed the AAKOMA protocol. The average time to attendance at the first session was approximately 3-4 weeks and during this intermediate time between completion of the protocol and initiation of treatment all patients were followed by study staff).
Time Frame: Post completion of 2 session Motivational Interviewing (MI) intervention (approximately 3-4 weeks on average during which time study staff followed all patients)
Measure: Number; unit: participants
Arm/Group | Motivational Interviewing Active | Delayed Control
Number analyzed (Participants) | 8 | 8
participants | 5 | 6

ADVERSE EVENTS:
Time Frame: Adverse event reporting occurred for the duration of data collection with this phase of the study from 2007 - 2011, including a 3 month follow up period after the last patient completed the protocol.
Description: Since the participants in the study were at-risk for depression or met criteria for depression and the purpose of the study was to assist the participants in securing treatment for their depression, we did not assess any of the patients as at risk for adverse events since they were being followed clinically by the study PI and the PI's mentors.
Arm/Group | Motivational Interviewing Active | Delayed Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
We lost 3 participants prior to intervention completion of the intervention which impacted results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No